CLINICAL TRIAL: NCT04240899
Title: Tele- Yoga for Adults With Anxiety: a Pilot Study
Brief Title: Yoga for Anxiety in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean-Francois Daneault, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # Pro2018002758
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease; Anxiety
Keywords: Yoga, anxiety, Parkinson's Disease, telerehabilitation
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a single group intervention study of adults (18-80 years-old) with Parkinson's Disease and anxiety symptoms undergoing a 6-week intervention of 30-minute yoga classes delivered remotely through videoconferencing 2-3 times per week. There will be baseline testing, a 6-week waiting period, timepoint-two testing, a 6-week intervention, post-intervention testing, and 6-week follow-up testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-yoga (Experimental): This is a single group study, therefore all subjects will be included in this single arm and will undergo the same telerehabilitation yoga intervention delivered through videoconferencing.
  Interventions: Other: Tele-yoga

INTERVENTIONS:
Other: Tele-yoga — Subjects will undergo 30-minute yoga sessions delivered remotely 2-3 times/week for 6-weeks. The yoga sessions will be delivered one-on-one and will include 5-7 minutes of breathing exercises 15-20 minutes of postures, and 5-7 minutes of relaxation and meditation exercises.

SUMMARY:
The purpose of this study is to investigate the effect of a telerehabilitation-yoga intervention delivered remotely via videoconferencing on adults with Parkinson's Disease and anxiety symptoms.

DETAILED DESCRIPTION:
A single group intervention study of adults (18-80 years-old) with Parkinson's Disease and anxiety symptoms undergoing a 6-week intervention of 30-minute yoga classes delivered remotely through videoconferencing 2-3 times per week. Subjects with symptoms of anxiety as indicated by their score on the Parkinson's Anxiety Scale will complete yoga classes delivered at-home with videoconferencing, receiving one-on-one yoga instruction including breathing, postures, and meditation/relaxation for two-three times a week. Data collection will occur remotely via videoconferencing at 0-weeks, 6-weeks after a waiting period, 12-weeks after the intervention, and 6-weeks after the last lab visit. Data collection will include demographics, mental health questionnaires, motor assessments, enjoyment, usability, and follow-up yoga status. Each yoga session will be video recorded to aide in recording adherence, adverse events, and challenges.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's Disease
* symptoms of anxiety as indicated by PAS (score ≥ 14)
* 18-80 years old
* ability to communicate verbally and follow directions
* English-speaking
* access to WiFi and applicable technological device (computer, laptop, tablet, smartphone etc.)
* willing to be video recorded during the yoga session
* willing to open Zoom on their technological device
* demonstrates self-reported technological literacy.

Exclusion Criteria:

* major depressive disorder (self-report medical history)
* injury or condition that could prevent engagement in yoga poses
* cognitive impairment or condition that would prevent the participant from understanding the tasks or communicating with the research team
* past yoga experience exceeding 5 or more times within the last 2 months
* pregnant women (self-report)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Parkinson's Anxiety Scale (PAS) | Baseline (at 0 weeks)
  The 12-item self-report PAS will be used to assess anxiety symptoms. It takes approximately 2-minutes to complete and is a 12-item scale with three sub-scales assessing 1. Persistent anxiety, episodic anxiety, and avoidance behavior. Participants answer questions on a scale from "not or never" (0) to "severe or almost always" (4) with a potential score range of 0-48. Higher score indicates greater symptoms of anxiety.
Parkinson's Anxiety Scale (PAS) | timepoint-2 (at 6-weeks)
  The 12-item self-report PAS will be used to assess anxiety symptoms. It takes approximately 2-minutes to complete and is a 12-item scale with three sub-scales assessing 1. Persistent anxiety, episodic anxiety, and avoidance behavior. Participants answer questions on a scale from "not or never" (0) to "severe or almost always" (4) with a potential score range of 0-48. Higher score indicates greater symptoms of anxiety.
Parkinson's Anxiety Scale (PAS) | post-intervention (at 12-weeks)
  The 12-item self-report PAS will be used to assess anxiety symptoms. It takes approximately 2-minutes to complete and is a 12-item scale with three sub-scales assessing 1. Persistent anxiety, episodic anxiety, and avoidance behavior. Participants answer questions on a scale from "not or never" (0) to "severe or almost always" (4) with a potential score range of 0-48. Higher score indicates greater symptoms of anxiety.
Parkinson's Anxiety Scale (PAS) | follow-up (at 18 weeks)
  The 12-item self-report PAS will be used to assess anxiety symptoms. It takes approximately 2-minutes to complete and is a 12-item scale with three sub-scales assessing 1. Persistent anxiety, episodic anxiety, and avoidance behavior. Participants answer questions on a scale from "not or never" (0) to "severe or almost always" (4) with a potential score range of 0-48. Higher score indicates greater symptoms of anxiety.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline (0 weeks), timepoint-2 (6-weeks), post-intervention (12-weeks) and at follow-up (6-weeks after post-intervention testing)
  The 21- item self-report BDI-II will be used to measure symptoms of depression. For each item the subject must choose one out of 4 statements of increasing severity regarding a specific symptom of depression. It is written approximately at a 5th grade reading level and takes about 5-10 minutes to complete. Potential scores range from 0-63 with higher scores indicating greater severity of depressive symptoms.
Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline (0 weeks), timepoint-2 (6-weeks), post-intervention (12-weeks) and at follow-up (6-weeks after post-intervention testing)
  The 50 item UPDRS will be used to assess motor and non-motor symptoms of Parkinson's Disease. It contains four sections 1. Mentation, Behavior, Mood; 2. Activities of Daily Living; 3. Motor Examination; and 4. Complications of Therapy. We will administer a modified version of this assessment in order to administer it remotely via videoconferencing. The hands on rigidity assessment will be excluded. Potential scores range from 0-179 (with rigidity components excluded), with higher scores indicating greater symptoms.
The Parkinson's Disease Questionnaire-39 (PDQ-39) | Baseline (0 weeks), timepoint-2 (6-weeks), post-intervention (12-weeks) and at follow-up (6-weeks after post-intervention testing)
  The 39-item self-report questionnaire will be used to asses quality of life. 8 domains (e.g. mobility, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort). It contains questions asking how often certain difficulties/problems have occurred within the last month with answers ranging from "never" to "always." Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty).
Five Times Sit to Stand Test (FTST) | Baseline (0 weeks), timepoint-2 (6-weeks), post-intervention (12-weeks) and at follow-up (6-weeks after post-intervention testing)
  The FTST, functional measure, will be administered to assess physical function. It will be administered using a chair in the participants' homes over a one-on-one Zoom videoconference. Participants will be encouraged to have another adult present during this portion of the data collection in case there is any loss of balance. Participants will be encouraged to use an armless chair approximately 63 centimeters from the ground and any deviation from this standard procedure will be documented. Time in seconds it takes the participant to raise from the chair 5 times will be recorded. Longer times will indicate poorer physical function.
Parkinson's Disease Sleep Scale-version 2 (PDSS-2) | Baseline (0 weeks), timepoint-2 (6-weeks), post-intervention (12-weeks) and at follow-up (6-weeks after post-intervention testing)
  The 15-item self report PDSS-2 measure will be used to assess sleep dysfunction. It contains questions about the participant's sleep experience during the past week with answers on a likert scale of 0-"very often" to 4-"never." Scores can range from 0-60 with higher scores indicating greater sleep impairment.
Adherence will be assessed by calculating the total number of yoga sessions attended. | Between week 6 to week 12
  Adherence to the yoga classes will be recorded each class including if a class is rescheduled. The occurrence, frequency, and brief description of any home yoga practice will also be recorded.
Adverse Events | Between week 6 to week 12
  All adverse events will be documented with a brief description of each adverse event, the potential relationship to the study, and the severity of each event.
Technical Difficulties Encountered | Between week 6 to week 12
  Anything perceived has a challenge by the yoga instructor or participant will be will be documented with severity of the challenge measured by time disrupted at an event level (time disrupted by the single event) and time disrupted from an entire session (time disrupted cumulatively).
Enjoyment/Feedback | Post-intervention testing (at 12-weeks)
  Enjoyment/feedback will be assessed via a Qualtrics questionnaire created by the study team inquiring about the subject's opinions about the intervention and a 10-point enjoyment scale.
Usability | Post-intervention testing (at 12-weeks)
  The systems usability scale, a 10-item scale that will be used to assess how usable the subjects feel that the tele-yoga intervention was. Scores are calculated such that a toal score of 100 is possible. Higher scores indicate higher usability.
Yoga Status at Follow-up | Follow-up (6-weeks after post-intervention)
  Yoga status at follow-up will be assessed via a Qualtrics questionnaire created by the study team asking questions about the subject's current involvement in yoga and other related topics.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Newark, New Jersey, United States

REFERENCES:
- [Derived] James-Palmer AM, Daneault JF. Tele-yoga for the management of Parkinson disease: A safety and feasibility trial. Digit Health. 2022 Aug 15;8:20552076221119327. doi: 10.1177/20552076221119327. eCollection 2022 Jan-Dec. PMID 35990111